CLINICAL TRIAL: NCT04561453
Title: A Prospective Feasibility Study of Multi-Platform Profiling Using Biospecimens From Patients With Resected Biliary Tract Cancer
Brief Title: Feasibility Study of Multi-Platform Profiling of Resected Biliary Tract Cancer
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to end of funding
Sponsor: University of Washington (Other)
Collaborators: Natera, Inc. (Industry); SEngine Precision Medicine, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: RG1121019; STUDY00010051 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder Cancer; Intrahepatic Cholangiocarcinoma; Perihilar Cholangiocarcinoma; Extrahepatic Cholangiocarcinoma; Hilar Cholangiocarcinoma; Distal Bile Duct Cancer
Keywords: organoid; circulating tumor DNA; ctDNA; drug screen; profiling; feasibility
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms; Klatskin Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resected Biliary Duct Cancer
  Interventions: Diagnostic Test: Multi-Platform Profiling with Organoid Drug Sensitivity Screening and ctDNA Monitoring

INTERVENTIONS:
Diagnostic Test: Multi-Platform Profiling with Organoid Drug Sensitivity Screening and ctDNA Monitoring — All patients in the study will have organoid creation and organoid drug sensitivity screening attempted on their fresh tumor tissue from surgical resection. All patients will also have blood taken pre-operatively and at multiple post-operative time points to monitor circulating tumor DNA.

SUMMARY:
This study is going to test the ability to successfully obtain results from certain personalized tests for patients with biliary tract cancers that are able to be surgically removed. Through surveys, this study will also evaluate the usefulness of these tests to medical oncologists as they make decisions on what standard or experimental treatments might benefit the patient's enrolled in the study. The study is observational and does not require any change in the standard approach to treating biliary tract cancer. Results of the personalized tests will be provided to the treating medical oncologist and the medical oncologist can choose to whether or not to change management based on these results. These personalized tests include reading of the cancer DNA, testing whether a panel of drugs can kill a patient's cancer cells in a test tube, and testing for small amounts of cancer DNA in the blood as a way to check for the presence of leftover cancer in the body after it is removed surgically. This study will also give extra pieces of cancer, that would otherwise be discarded, from surgery for laboratory research into how biliary tract cancers respond to drugs and the body's immune system. The investigators hypothesize that the drug screen test will, in some cases, be useful to the medical oncologist and may lead to the use of cancer drugs that would not otherwise have been chosen based on standard guidelines or based on cancer DNA testing. The investigators hypothesize that the test tube drug screening method will correlate with how the cancer responds to the drugs in real life for those patients that end up receiving a drug that was included in the drug screen panel. The investigators hypothesize that monitoring of cancer DNA in the blood stream will help us predict which patients are most likely to have their cancer return after surgery. The investigators also hypothesize that in many cases the appearance of cancer DNA in the blood stream will happen weeks to months prior to the cancer showing up on usual body imaging or other lab tests. Finally, the investigators hypothesize that, for patients undergoing medical treatment for their cancer, trends in the amount of cancer DNA in the blood stream will correlate with the effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in the study:

* Be ≥18 years of age.
* Have a preoperative biopsy with a histopathological diagnosis consistent with a biliary tract cancer (intrahepatic or extrahepatic cholangiocarcinoma or gallbladder carcinoma) or, absent a biopsy, have a clinical presentation consistent with a biliary tract cancer, and are eligible for curative resection
* Surgical candidate for the requisite resection as assessed by a liver surgeon or as assessed by, if deemed necessary, a pre-operative evaluation by internal medicine, cardiology and/or anesthesia.
* Pre-operative imaging showing a measurable amount of disease that, per the judgement of the surgical oncologist, will be enough to allocate to at least genomic profiling as well as the organoid creation portion of this research study.
* Be willing to undergo surgical resection and willing to have the surgery performed at University of Washington.
* Be willing to follow-up with medical oncology post-operatively and allow the study team to collect longitudinal data on their course as well as longitudinal blood samples for circulating tumor DNA surveillance
* Have an ECOG performance status of 0-2.
* Have an expected survival of ≥6 months.
* Have adequate bone marrow function as evidenced by:

  1. Absolute neutrophil count ≥1,000/mm3 or 1.0 ×10^9/L
  2. Hemoglobin ≥8 g/dL
  3. Platelets ≥60,000/mm3 or 60 × 10^9/L
* Have adequate hepatic function as evidenced by the below, or are expected to have adequate hepatic function (as defined below) post-operatively:

  1. Serum total bilirubin ≤2 × upper limit of normal (ULN), unless considered due to Gilbert's disease or a biliary obstruction
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤8 × ULN
* Have adequate renal function as evidenced by the below or are expected to have adequate renal function (as defined below) post-operatively:

  a. Serum creatinine <1.5 × ULN OR b. Creatinine clearance ≥50 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR) estimation: (140 - Age) x (weight in kg) x (0.85 if female)/72 x sCr
* Be able to understand and willing to sign the informed consent form and to comply with scheduled visits, treatment plans, procedures, and laboratory tests, including serial peripheral blood sampling, during the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled in the study:

* Mixed hepatocellular carcinoma-cholangiocarcinoma on histology.
* Refuses to sign the consent.
* Received any prior systemic targeted therapy (excludes chemotherapy) or an investigational agent directed at their presumed cholangiocarcinoma prior to resection
* Received any prior radiation or catheter-directed therapy to the malignant tumor being resected, unless there has been definitive malignant progression of that tumor since the time of the post-treatment imaging assessment after radiation or catheter-directed therapy.
* Received any systemic anticancer therapy or an investigational agent for another indication (a synchronous cancer of a different primary site) in the 6 months prior to discovery of their presumed cholangiocarcinoma by imaging
* Have known extrahepatic metastases or locally advanced disease precluding resection of the cholangiocarcinoma.
* Have a history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid or liquid tumor with no known active disease present that, in the opinion of the Investigator, will not affect subject outcome in the setting of current cholangiocarcinoma diagnosis.
* Are pregnant or breastfeeding
* Have any other acute or chronic medical or psychiatric condition, including recent (within 12 months of cholangiocarcinoma diagnosis) or active suicidal ideation or behavior, or a laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
* Have been committed to an institution by virtue of an order issued either by the judicial or administrative authorities.
* Are dependent on the Sponsor, Investigator, or study site, per local institution regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from a group of individuals being evaluated at University of Washington and the Seattle Cancer Care Alliance for a liver mass that is suspected to be localized biliary tract cancer amenable to resection.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Success Rate of Organoid Culture and Drug Screen | Within 12 weeks after surgery
  The investigators will measure the percentage of patients for whom organoids are able to be successfully cultured and subjected to a drug screen.
Success Rate of Obtaining circulating tumor DNA (ctDNA) quantification and Ability to assess change in ctDNA levels across those time points | Through study completion, an average of 4 years.
  The investigators will measure the percentage of patients for whom ctDNA was able to be collected and quantified at multiple key time points across the course of a patient's treatment.

SECONDARY OUTCOMES:
Physician-Adjudicated Utility of Profiling Test Results - Post-Adjuvant Therapy | At the time of completion of adjuvant therapy, on average 6 months after surgery.
  Through surveys, the investigators will ask cancer physicians how helpful the profiling test results are anticipated to be to the ultimate management of the patient after they have received adjuvant chemotherapy.
Prospective Concordance of Organoid Drug Screen Results and In Vivo Drug Activity | Through study completion, an average of 4 years.
  For patients that are treated with drugs that were also evaluated by the initial organoid drug screen, the investigators will measure how often the organoid's response to the drug paralleled the response of the cancer to the drug when administered to the patient.
Predictive Value of circulating tumor DNA (ctDNA) for Recurrence | From date of randomization until the date of first documented radiographic recurrence, an average of 2 years after surgery.
  The investigators will evaluate how often measurable post-operative ctDNA levels were able to predict ultimate recurrence of clinical disease. The investigators will measure the lead time of ctDNA-assessed recurrence over radiographic recurrence.
Concordance of Organoid Drug Screen Results with Next Generation Sequencing (NGS)-Predicted Drug Sensitivities | Within 12 weeks after surgery when results of NGS and Organoid Drug Screen have returned.
  The investigators will evaluate how often the organoid drug screen responded to a drug that genomic profiling by NGS would have predicted the cancer would be sensitive to.
Physician-Adjudicated Utility of Profiling Test Results - At Time of Recurrence | At the time of cancer recurrence, on average 24 months after surgery.
  Through surveys, the investigators will ask cancer physicians how helpful the profiling test results were to the ultimate management of the patient at the time their cancer recurred.
Predictive Value of circulating tumor DNA (ctDNA) for Response to Medical Therapy | Through study completion, an average of 4 years.
  The investigators will correlate ctDNA level trends with radiographic responses to medical treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gentry King, MD, Principal Investigator — University of Washington Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No